CLINICAL TRIAL: NCT03270891
Title: Determining the Feasibility, Acceptability, and Preliminary Effectiveness of Pharmacogenomic Testing in Primary Care
Brief Title: Pharmacogenomic Testing in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Lorraine Buis, Assistant Professor, Family Medicine Assistant Professor of Information, School of Information, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00121185
Record Dates: First submitted 2017-08-28; First posted 2017-09-01 (Actual); Results first posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Antidepressants Causing Adverse Effects in Therapeutic Use
Keywords: Pharmacogenomics; Primary care physicians
MeSH Terms: interventions — Pharmacogenomic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Delayed intervention (control arm) (Active Comparator): Patients in this arm will have PGx test results made available to physicians 3 months after study enrollment
  Interventions: Diagnostic Test: PGx test
- PGx Test (Experimental): Patients in this arm will have PGx test results made available to physicians as soon available after enrollment.
  Interventions: Diagnostic Test: PGx test

INTERVENTIONS:
Diagnostic Test: PGx test — A laboratory developed genetic test that differentiates common and uncommon alleles in genes that have been previously identified as being involved in either the metabolism or response of drugs used in the treatment of depression and/or anxiety. The results are provided as a report that contains information related to the allele status of the patient's genes, translates this into a phenotype, and relates this phenotype to recommendation classes for drugs.
  Other Names: Pharmacogenomic test; Progenity Informed PGx test

SUMMARY:
This is a 6-month randomized, wait-listed, controlled pilot trial conducted in 6 department of family medicine (DFM) clinics at the University of Michigan (UM). Physicians practicing at a UM DFM clinical site who are willing to utilize pharmacogenomic (PGx) test results to manage antidepressant use will be enrolled. Patients of these DFM physicians who are adults with a new prescription for a target antidepressant will also be enrolled.

DETAILED DESCRIPTION:
This is a 6-month randomized, wait-listed, controlled pilot trial conducted in 6 department of family medicine (DFM) clinics at the University of Michigan (UM). We will enroll physicians practicing at a UM DFM clinical site who are willing to utilize PGx test results in conjunction with treating patients prescribed certain antidepressants. We will also enroll patients of these DFM physicians who are adults with a new prescription for an antidepressant (within the past 4 weeks) including patients who have switched to a new antidepressant from another antidepressant or have added on a new antidepressant to current antidepressant therapy. Patients are excluded if taking an antidepressant for more than 4 weeks or if they have had PGx testing in the past. Patients will be randomized to either an intervention or control group. Patients in the intervention group will have PGx test results available soon after enrollment while the control patients will have test results available 3 months after the first visit. All patients will complete a baseline, 3-, and 6-month assessment; control patients will have an additional 9-month assessment. Data to be collected include symptoms and severity (PHQ-8, GAD7), functional health status (SF-12), PGx knowledge, work status changes, demographic information, physician and emergency department visits, adverse effects, and medication alterations and adherence.

ELIGIBILITY:
Physician participants

Inclusion criteria:

* Be a practicing physician at a University of Michigan Department of Family Medicine clinic
* Be willing to use PGx test results for their patients enrolled in the study
* Be willing to allow study staff to contact their patients
* Self-report that they are willing to prescribe antidepressants

Exclusion criteria:

-Do not meet inclusion criteria

Patient Participants

Inclusion:

* Be a patient of a participating physician
* Have a new prescription for one of the following antidepressant medications: citalopram (Celexa), escitalopram (Lexapro), fluoxetine (Prozac, Prozac Weekly, Rapiflux, Sarafem, Selfemra), fluvoxamine (Luvox, Luvox CR), paroxetine (Paxil, Paxil CR), sertraline (Zoloft), duloxetine (Cymbalta, Irenka), venlafaxine (Effexor), venlafaxine XR (Effexor XR), nortriptyline (Aventyl, Pamelor), bupropion (Forfivo XL, Wellbutrin, Wellbutrin SR, Wellbutrin XL), mirtazapine (Remeron, Remeron Soltab), or vortioxetine (Trintellix)
* Be willing to undergo PGx testing via single tube blood draw

Exclusion:

* Do not speak English
* Have previously undergone PGx testing
* Are unable to provide their own consent to participate in the study
* Have been taking the new antidepressant prescription for longer than 4 weeks (prior to screening)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2021-09-05 (Actual); Study Completion 2022-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorriane Buis, PhD, Principal Investigator — University of Michigan Department of Family Medicine
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Manzor Mitrzyk B, Kadri R, Farris KB, Ellingrod VL, Klinkman MS, Ruffin Iv MT, Plegue MA, Buis LR. Using Pharmacogenomic Testing in Primary Care: Protocol for a Pilot Randomized Controlled Study. JMIR Res Protoc. 2019 Aug 19;8(8):e13848. doi: 10.2196/13848. PMID 31429417

RESULTS

PARTICIPANT FLOW:
Groups:
- Physicians: Physicians who practiced at 1 of the 6 UM Family Medicine clinics.
Period: Overall Study
Arm/Group | Delayed Intervention (Control Arm) | PGx Test | Physicians
Started | 26 | 25 | 24
Received Intervention | 25 | 25 | 0
For Physician Arm Only; Those Physicians Who Had Patients Who Participated | 0 | 0 | 17
Completed | 22 | 19 | 17
Not Completed | 4 | 6 | 7
Not completed — Lost to Follow-up | 3 | 6 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — For Physician arm only; those physicians who did not have patients who participated | 0 | 0 | 7

BASELINE CHARACTERISTICS:
Population: 1 participant was withdrawn by the study staff and PI after baseline data was collected but before receiving the intervention.
Groups:
- Delayed Intervention (Control Arm): Participants in this arm will have PGx test results made available to physicians 3 months after study enrollment
  PGx test: A laboratory developed genetic test that differentiates common and uncommon alleles in genes that have been previously identified as being involved in either the metabolism or response of drugs used in the treatment of depression and/or anxiety. The results are provided as a report that contains information related to the allele status of the patient's genes, translates this into a phenotype, and relates this phenotype to recommendation classes for drugs.
- PGx Test: Participants in this arm will have PGx test results made available to physicians as soon available after enrollment.
  PGx test: A laboratory developed genetic test that differentiates common and uncommon alleles in genes that have been previously identified as being involved in either the metabolism or response of drugs used in the treatment of depression and/or anxiety. The results are provided as a report that contains information related to the allele status of the patient's genes, translates this into a phenotype, and relates this phenotype to recommendation classes for drugs.
- Total: Total of all reporting groups
Arm/Group | Delayed Intervention (Control Arm) | PGx Test | Physicians | Total
Number analyzed (Participants) | 26 | 25 | 24 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Physician age is reported as a study specific outcome measure so that the total means are not mixed between participants and physicians.
  years
    number analyzed (Participants) | 26 | 25 | 0 | 51
    (all) | 39.2 (13.2) | 42.0 (14.6) |  | 40.5 (13.9)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 13 | 10 | 8 | 31
  Female | 13 | 14 | 16 | 43
  Other | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 23 | 19 | 19 | 61
  Black | 1 | 1 | 0 | 2
  Asian | 1 | 1 | 3 | 5
  Other | 0 | 2 | 2 | 4
  Unknown | 1 | 2 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 25 | 24 | 75
Marital Status [Count of Participants; unit: Participants] — Population: Protocol had no plans to collect marital status from physicians.
  Participants
    Not Married: number analyzed (Participants) | 26 | 25 | 0 | 51
    Not Married | 15 | 10 |  | 25
    Married: number analyzed (Participants) | 26 | 25 | 0 | 51
    Married | 11 | 15 |  | 26
Education [Count of Participants; unit: Participants]
  <4 yrs College | 8 | 11 | 0 | 19
  Bachelor's Degree | 7 | 6 | 0 | 13
  Graduate | 11 | 8 | 24 | 43
Employment [Count of Participants; unit: Participants]
  Unemployed | 7 | 8 | 0 | 15
  Employed | 19 | 17 | 24 | 60
Income [Count of Participants; unit: Participants] — Population: Protocol had no plans to collect income status from physicians.
  Participants
    <50k: number analyzed (Participants) | 26 | 25 | 0 | 51
    <50k | 7 | 8 |  | 15
    50k-99k: number analyzed (Participants) | 26 | 25 | 0 | 51
    50k-99k | 10 | 7 |  | 17
    100k+: number analyzed (Participants) | 26 | 25 | 0 | 51
    100k+ | 9 | 10 |  | 19
Number of Children [Count of Participants; unit: Participants] — Population: Protocol had no plans to collect number of children data from physicians.
  Participants
    No Children: number analyzed (Participants) | 26 | 25 | 0 | 51
    No Children | 14 | 13 |  | 27
    At Least One: number analyzed (Participants) | 26 | 25 | 0 | 51
    At Least One | 12 | 12 |  | 24
Smoking Status [Count of Participants; unit: Participants] — Population: Protocol had no plans to collect smoking status from physicians.
  Participants
    Non-Smoker: number analyzed (Participants) | 26 | 25 | 0 | 51
    Non-Smoker | 25 | 23 |  | 48
    Smoker: number analyzed (Participants) | 26 | 25 | 0 | 51
    Smoker | 1 | 2 |  | 3
Age of Physicians, Continuous [Mean (Standard Deviation); unit: years] — Population: This measure is for physician age only so it does not include patient participant data, in order to have the patient participant data mean totals remain accurate. Therefore patient participants are not analyzed here.
  years
    number analyzed (Participants) | 0 | 0 | 24 | 24
    (all) |  |  | 41.83 (10.47) | 41.83 (10.47)

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants Prescribed Antidepressant Medication
Description: Count of participants who have been prescribed antidepressant medications which are not contraindicated
Time Frame: Baseline, 3 months, 6 months, and 9 months
Population: Per protocol, only control arm patients were to have a 9 month assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Delayed Intervention (Control Arm) | PGx Test
Number analyzed (Participants) | 25 | 25
Participants
  Baseline | 5 | 8
  Month 3 | 5 | 8
  Month 6 | 6 | 8
  Month 9: number analyzed (Participants) | 25 | 0
  Month 9 | 5 |

2. Secondary Outcome: Change in Symptom Severity - Patient Health Questionnaire (PHQ-8)
Description: Change in PHQ-8 scores. The PHQ-8 is an 8-item participant-report measure for screening for depression and for establishing depression severity. The total score ranges from 0-24, with a higher score indicating greater depression symptom severity.
Time Frame: Baseline and 6 months
Population: PHQ-8 data is unavailable for 8 participants in the control arm and 7 participants in the PGx Test arm because of missing data at 6 months or loss to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Delayed Intervention (Control Arm) | PGx Test
Number analyzed (Participants) | 25 | 25
score on a scale
  Baseline | 9.0 (4.4) | 8.6 (6.1)
  6 month: number analyzed (Participants) | 17 | 18
  6 month | 7.5 (4.3) | 5.8 (5.4)
Statistical Analysis 1: Comparison: Delayed Intervention (Control Arm); Baseline and 6 month values; Test type: Superiority — Null hypothesis of equality; p = 0.0115, t-test, 2 sided
Statistical Analysis 2: Comparison: PGx Test; baseline to 6 month comparison; Test type: Superiority — Null hypothesis of equality; p = 0.027, t-test, 2 sided

3. Secondary Outcome: Change in Symptom Severity - General Anxiety Disorder - 7 (GAD 7)
Description: The GAD-7 is a self-administered assessment for general anxiety disorder. The total score for the seven items ranges from 0 to 21. Higher values represent a worse outcome.
Time Frame: Baseline and 6 months
Population: Because GAD-7 data is unavailable for 8 participants in the control arm and 7 participants in the PGx Test arm because of missing data at 6 months or loss to follow-up, the data is presented for those participants who had both data points so comparisons between the two time points are appropriate.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Delayed Intervention (Control Arm) | PGx Test
Number analyzed (Participants) | 17 | 18
score on a scale
  baseline | 9.1 (6.2) | 6.9 (5.6)
  Month 6 | 6.1 (5.0) | 5.2 (4.9)
Statistical Analysis 1: Comparison: Delayed Intervention (Control Arm); Baseline p value to six month; Test type: Superiority — Null hypothesis of equality; p = 0.0327, t-test, 2 sided
Statistical Analysis 2: Comparison: PGx Test; baseline to 6 month comparison p value; Test type: Superiority — Null hypothesis of equality; p = 0.2088, t-test, 2 sided

4. Secondary Outcome: Change in Adherence to Refills and Medication Scale (ARMS) Scores
Description: Change in medication adherence: The Adherence to Refills and Medication was scored by summing together the 14 items after first reversing the final item to be consistent in direction with the others. Individuals were allowed to have up to 2 missing values present which were imputed with the mean of the remaining answered items, only a handful of individuals answered 13 of the 14 questions resulting in a single item within their scale being imputed across the time periods.
  The questionnaire has 14 items with each item being recorded on a four-point Likert scale. The total score ranges from 14-56 with the lower score indicating better adherence.
Time Frame: Baseline and 6 months
Population: ARMs data is unavailable for 10 participants in the control arm and 8 participants in the PGx Test arm because of missing data at 6 months or loss to follow-up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Delayed Intervention (Control Arm) | PGx Test
Number analyzed (Participants) | 15 | 17
score on a scale
  baseline | 17.1 (3.3) | 17.4 (3.2)
  6 month | 17 (2.5) | 16.6 (3.2)
Statistical Analysis 1: Comparison: Delayed Intervention (Control Arm); baseline to 6 month comparison; Test type: Superiority — Null hypothesis of equality; p = 0.947, t-test, 2 sided

5. Other Pre Specified Outcome: Acceptability of PGx Testing
Description: Acceptability of PGx testing in primary care among persons taking a target antidepressant and primary care physicians who care for them
Time Frame: Baseline and 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: six months
Description: Per protocol and because they received no intervention, no adverse event data was intended to be collected from physicians, so they are not presented here.
Arm/Group | Delayed Intervention (Control Arm) | PGx Test
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25
Other Adverse Events (participants affected / at risk) | 0/26 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT03270891/Prot_SAP_000.pdf